CLINICAL TRIAL: NCT06462469
Title: A Single-arm, Multi-center Study of Ruxolitinib for the Treatment of Chinese Patients With Grade II-IV Corticosteroid-refractory Acute Graft Versus Host Disease
Brief Title: Study of Efficacy and Safety of Ruxolitinib in Patients With Grade II to IV Steroid-refractory Acute Graft vs. Host Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424C2416
Record Dates: First submitted 2024-06-05; First posted 2024-06-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Steroid-refractory Acute Graft Versus Host Disease
Keywords: SR-aGvHD; aGvHD; acute graft-versus-host disease; ruxolitinib; Chinese patients; corticosteroid-refractory; Grade II-IV; Grade II to IV
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Participants will receive ruxolitinib orally of 10 mg BID daily (given as two 5-mg tablets, approximately 12 hours apart).
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is taken orally daily at 10 mg BID, given as two 5-mg tablets.
  Other Names: INC424

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ruxolitinib therapy in Chinese adults and adolescents (≥ 12 years old) with Grade II-IV steroid-refractory acute graft versus host disease (SR-aGvHD).

DETAILED DESCRIPTION:
Participants will start with a screening period to assess the eligibility; only participants who meet all the inclusion and none of the exclusion criteria will start study treatment from Day 1 to Week 24 or end of treatment. Following safety follow up visits, participants will receive the long-term follow-up until Month 12.

ELIGIBILITY:
Key Inclusion criteria

* Male or female Chinese participants aged 12 or older at the time of informed consent. Written informed consent from participant, parent or legal guardian.
* Able to swallow tablets.
* Have undergone alloSCT from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood.
* Clinically diagnosed Grades II to IV acute GvHD as per standard criteria occurring after alloSCT requiring systemic immune suppressive therapy.
* Evident myeloid and platelet engraftment (confirmed within 48 hours prior to study treatment (ruxolitinib) start):
* Confirmed diagnosis of steroid refractory aGvHD defined as participants administered systemic corticosteroids (methylprednisolone at least 1 mg/kg/day [or equivalent prednisone dose at least 1.25 mg/kg/day]), given alone or combined with calcineurin inhibitors (CNI) and either:

  1. Progression based on organ assessment after at least 3 days compared to organ stage at the time of initiation of systemic corticosteroid +/- CNI for the treatment of Grade II to IV aGvHD. OR
  2. Failure to achieve at a minimum partial response based on organ assessment after 7 days compared to organ stage at the time of initiation of systemic corticosteroid +/-CNI for the treatment of Grade II to IV. OR
  3. Participants who fail corticosteroid taper defined as fulfilling either one of the following criteria:

     * Requirement for an increase in the corticosteroid dose to methylprednisolone ≥ 1 mg/kg/day (or equivalent prednisone dose ≥ 1.25 mg/kg/day). OR
     * Failure to taper the methylprednisolone dose to < 0.5 mg/kg/day (or equivalent prednisone dose <0.6 mg/kg/day) for a minimum of 7 days.

Key Exclusion criteria

* Has received more than one systemic treatment for steroid refractory aGvHD. Participants who received JAK inhibitor therapy for any indication after initiation of current alloSCT conditioning.
* Clinical presentation resembling de novo chronic GvHD or GvHD overlap syndrome with both acute and chronic GvHD features.
* Failed prior alloSCT within the past 6 months. Presence of relapsed primary malignancy after the alloSCT was performed.
* Presence of an active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment.
* SR-aGvHD occurring after non-scheduled donor lymphocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence. Note: Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
* Presence of significant respiratory disease, severely impaired renal function, clinically significant or uncontrolled cardiac disease, unresolved cholestatic and liver disorders (not attributable to aGvHD). Disorders and/or current therapy with medications that interfere with coagulation or platelet function.

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2028-02-17 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Day 28 per Investigators | Day 28
  The ORR at Day 28 defined as the percentage of participants demonstrating a complete response (CR) or partial response (PR) without requirement for additional systemic therapies for an earlier progression, mixed response or nonresponse, according to standard criteria and assessed by investigators.

SECONDARY OUTCOMES:
Durable Overall response rate (ORR) at Day 56 | Day 56
  Durable ORR at Day 56 is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) at Day 28 and maintain a CR or PR at Day 56.
Duration of Response (DOR) | From Week 1 to long term follow up Month 12
  DOR is defined as the time from first response until aGvHD progression or the date of additional systemic therapies for aGvHD.
Best overall response (BOR) | From week 1 to Day 28
  Percentage of participants who achieved overall response (complete response (CR) + Partial response (PR) at any time point up to and including Day 28 and before the start of additional systemic therapy for aGvHD.
Overall survival (OS) | From the date of start of study treatment to date of death, up to approx. 12 months
  Overall survival (OS) is defined as the time from the date of start of study treatment to date of death due to any cause.
Non-relapse mortality (NRM) | From date of start of study treatment to date of death, up to approx. 12 months
  Non-relapse mortality (NRM) is defined as the time from date of start of study treatment to date of death not preceded by hematologic disease relapse/progression.
Event-free survival (EFS) | From the date of start of study treatment to the date of hematologic disease relapse/progression, graft failure, or death, up to approx. 12 months
  Event-free survival (EFS) is defined as the time from the date of start of study treatment to the date of hematologic disease relapse/progression, graft failure, or death due to any cause.
Failure-free survival (FFS) | From the date of start of study treatment to date of hematologic disease relapse/progression, non-relapse mortality, or addition of new systemic aGvHD treatment, up to approx. 12 months
  Failure-free survival (FFS) is defined as the time from the date of start of study treatment to date of hematologic disease relapse/progression, non-relapse mortality, or addition of new systemic aGvHD treatment.
Malignancy Relapse/Progression (MR) | From date of start of study treatment to hematologic malignancy relapse/progression, up to approx. 12 months
  Malignancy Relapse/Progression (MR) is defined as the time from date of start of study treatment to hematologic malignancy relapse/progression. Calculated for participants with underlying hematologic malignant disease.
Reduction of daily corticosteroids dose | Up to Day 56
  This includes the assessment of systemic corticosteroid use and daily dose, and the percentage of participants successfully tapered off all systemic corticosteroids until Day 56, by time intervals and overall.
Cumulative incidence of chronic GvHD | From Week 1 to long term follow up of month 12
  Cumulative incidence of chronic GvHD (cGvHD) includes mild, moderate and severe occurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- China (13):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Taian
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com